CLINICAL TRIAL: NCT06935812
Title: Comparison of the Effects of Bimanual, Finger and Virtual Reality Exercises in Individuals With Mild Cognitive Impairment - Randomized Controlled Study
Brief Title: Comparison of the Effects of Bimanual, Finger and VR Exercises in PwMCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Betül Fatma Bilgin, Research Assistant, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETK00-2024-0113
Record Dates: First submitted 2024-06-01; First posted 2025-04-20 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Finger Exercise; Bimanual Exercise; Virtual Reality; Processing Speed; Cognitive Functions; Walking Speed; Gross Motor Skills; Fine Motor Skills; Dual Task
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bimanual Exercise (Experimental): Bimanual Exercise The bimanual exercise group consists of exercises that involve movements in which both hands are used simultaneously. The bimanual exercise group will have 40 minutes of training for 3 sessions per week for 8 weeks.
  Interventions: Other: Bimanual Exercise
- Finger Exercise (Experimental): Finger Exercise The finger exercise group consists of exercises that involve finger movements. The bimanual exercise group will have 40 minutes of training for 3 sessions per week for 8 weeks.
  Interventions: Other: Finger Exercise
- Virtual Reality (Experimental): Virtual Reality The virtual reality exercise group consists of hand-tracking game exercises that involve finger movements. The bimanual exercise group will have 40 minutes of training for 3 sessions per week for 8 weeks.
  Interventions: Other: Virtual Reality
- Control (No Intervention): In this group, participants will asses on the first and the last weeks of the program (0. and 8. week).

INTERVENTIONS:
Other: Bimanual Exercise — The bimanual exercise group consists of exercises that involve movements in which both hands are used simultaneously. The bimanual exercise group will have 40 minutes of training for 3 sessions per week for 8 weeks.
  Arms: Bimanual Exercise
Other: Finger Exercise — The finger exercise group consists of exercises that involve finger movements. The bimanual exercise group will have 40 minutes of training for 3 sessions per week for 8 weeks.
  Arms: Finger Exercise
Other: Virtual Reality — The virtual reality exercise group consists of hand-tracking game exercises that involve finger movements. The bimanual exercise group will have 40 minutes of training for 3 sessions per week for 8 weeks.
  Arms: Virtual Reality

SUMMARY:
Mild Cognitive Impairment (MCI) is defined as an impairment in a single cognitive function, usually memory, other than normal cognitive decline with age, that does not fulfil dementia criteria. Finger movements have been shown to stimulate the sensory-motor and cognitive parts of the cerebral cortex, as well as the supplementary motor area, Broca's area, premotor cortex, and prefrontal cortex, all of which contribute to movement skills. Asymmetrical hand and finger movements done concurrently were proven to improve cognitive processes and cerebral blood flow more than movements performed with one hand.

DETAILED DESCRIPTION:
Cognitive impairment is one of the most pressing healthcare problems of the 21st century. Mild cognitive impairment (MCI) has been defined as a disorder in a single cognitive function; usually, memory is impaired to an extent greater than anticipated for age, yet the patient does not meet the criteria for dementia. MCI, known as a risk factor for the early stage of dementia, constitutes a risk factor for Alzheimer's Disease (AD) and is also known as the prodromal syndrome of AD. MCI affects 3%-22% of people over the age of 65, depending on demographic characteristics, and persons with MCI (PwMCI) progress to dementia at a rate of 10%-15% every year. Advanced age, low education level, and low cognitive capacity are among the most common risk factors for MCI. Although the pathology of MCI is not completely understood, hippocampal and entorhinal cortex atrophy is defined as a hallmark, and the connectivity of the hippocampus with the prefrontal lobe, temporal lobe, parietal lobe, and cerebellum was found to be lower in PwMCI than healthy controls. PwMCI can be categorized as amnestic and non-amnestic MCI. Individuals with non-amnestic MCI have impairments in other domains than memory, such as attention/executive functions (eMCI), which are frequent and disabling symptoms MCI. It was shown that response inhibition, switching, and cognitive flexibility are selectively impaired, while sustained and divided attention are intact in PwMCI. It has been proposed that executive control and gait share common frontal brain circuitry vulnerable to age-related neuropathology. It is known that cognitive deficits are associated with increased fall risk in community-dwelling older adults, and older adults with higher cognitive impairments are more prone to experience falls. The stepping reaction time variability indicate compromised neural circuitry involved in executive function, gait, and posture and increases the risk of fall in PwMCI.

A promising avenue in this regard is finger or hand exercise, which is rooted in traditional Chinese medicine and grounded in the meridian theory. The meridian theory suggests that specific meridians and acupoints can be stimulated through finger exercises, leading to the promotion of energy flow and restoration of overall balance within the body. While finger exercise has a historical foundation in traditional Chinese medicine, its potential impact on cognitive function has recently gained attention, resulting in several studies investigating its benefits. Notably, two recent randomized controlled trials (RCT) demonstrated that finger exercise improved cognitive performance in both cerebral ischemic stroke (CIS) and mild cognitive impairment (MCI) patients. Despite the promising nature of finger exercises as an effective cognitive intervention highly accessible to older adults, a thorough investigation of their effects is imperative before widespread application.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are between 50-75 years of age
* Individuals diagnosed with MCI by a geriatrician according to DSM-5 criteria,
* Who has the Montreal Cognitive Assessment score between 13-26,
* Who has the Quick Mild Cognitive Impairment screen score between 48-67,
* Who has Instrumental Activities of Daily Living Scale score ≥6/8,
* Who says yes to "Do you have a memory problem?" question,
* Who can walk independently without using any walking aids

Exclusion Criteria:

* Participants who have any musculoskeletal disorders that may cause balance and gait disorders,
* Who have central or peripheral neurological diseases (eg. stroke, Parkinson's disease or polyneuropathies),
* Who are using psychiatric drugs that may affect psychiatric disease and/or cognitive performance (Using nonsteroidal anti-inflammatory drugs more than three times a week, which may affect cognitive functions, using gingko biloba and antioxidant supplements (for example, coenzyme Q10 and alpha-lipoic acid)),
* Who has daltonism and
* Who attends any exercise program last 6 months will not be included in this study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
MoCA | 8 weeks
  Montreal Cognitive Assessment Scale: MoCA is a short screening test for Mild Cognitive Impairment and Alzheimer's Disease to measure cognitive functions. The test is administered using pen and paper and takes approximately 10-20 minutes. It has 7 subheadings and these are listed as follows: (1) visuospatial/executive functions (clock drawing and cube copying, tracing test (part B) - 5 points); (2) naming (learning and repeating a list of 5 words - 3 points); (3) memory (5 points for recall); (4) attention (target-orientated clapping - 6 points); (5) language (fluency - 3 points); (6) abstract thinking (similarity between words - 2 points); and (7) orientation (knowledge of day, month, year and place - 6 points). The score range is 0 to 30, with higher scores indicating better performance. Values below 26 points indicate a risk of cognitive impairment and provide information about a possible MCI.
Cognitive functions-Trail Making Test (A-B) | 8 weeks
  Trail Making Test (A-B): Trail Making Test (TMT) is a complex visual screening test with motor components and is sensitive to frontal region functions (12, 13). Motor speed, agility and careful participation are required to be successful in this test. This first version of the IST consists of two parts (forms), A and B. In Part A, the participants will be asked to connect the circles with numbers (1-2-3-4-......) on the test form by drawing a line consecutively and in the correct order. In Part B, the participants will be asked to connect the circles containing numbers and letters (1-A,2-B,3-C- ......) on the test form by drawing a line in a consecutive and correct order in accordance with the order of one number and one letter. The time will be recorded for both A and B tests.
Cognitive functions-Digit Span Test/Digit Symbol Substitution Test | 8 weeks
  Digit Span Test (DST): In the DST, participants will be asked to repeat the read digits in sequence. The test continues with growing digits. Then, in the second part of the test, they will be asked to repeat the spoken digits backwards and the number of correct ones will be recorded.
  Digit Symbol Substitution Test (DSST): DSST is a test used to evaluate psychomotor performance. The participants will be asked to draw the symbol determined for each number in the boxes left blank for 90 seconds. The total number of correct shapes will be recorded.
Cognitive Functions-Verbal Fluency Test/Serial Subtraction Test | 8 weeks
  Verbal Fluency Test - Phonemic: The participant is asked to count the words starting with the letters we have determined (letters A and S) within 1 minute. The number of correct and incorrect words spoken will be determined.
  Serial Subtraction Test: The participant is asked to count backwards by subtracting 7 from a number between 200-300 within 1 minute. The number of correct and incorrect counts will be determined.

SECONDARY OUTCOMES:
Choice Stepping Reaction Time Mat (CSRT) | 8 weeks
  Lower extremity reaction time: Step taking reaction time will be evaluated on the Choice Stepping Reaction Time Mat (CSRT) with Flash/response facilitation (stepping as fast as possible in the direction of the lit green arrow) and Inhibitor/response inhibition (staying in place when the purple arrow is lit and stepping with the green arrow). Accordingly, reaction time, movement time and response/operation time (sum of reaction time and movement time) will be evaluated in all tests.
  Upper extremity reaction time:
  While the participant is in a sitting position, he/she will be asked to touch the buttons (Blaze Pods) on the table as fast as possible when the light is on and the reaction time will be recorded. The test will be performed separately for right and left extremities.

OTHER OUTCOMES:
Grip Strength | 8 weeks
  Hand held dynamometer: A hand held dynamometer will be used to measure grip strength, which begins to decline with ageing. The participant will sit with the shoulder in adduction, elbow in 90 degree flexion, forearm and wrist in neutral position. The therapist will then place the dynamometer in the hand of the person being tested and ask them to squeeze as hard as possible. The participants will be asked to grasp the grip with all their strength for both hands and the average of the three repetitions will be taken.
Fine motor skills | 8 weeks
  Purdue Pegboard Test:
  The total duration of the test, including the introduction time, is 5-10 minutes. The materials required are a rectangular pegboard with 25 holes along two rows and a stopwatch. At the end of the application, a total of five different scores will be obtained with measurements such as right hand, left hand, both hands together, combined task and sum of scores. During the application, the person will be asked to insert the nails into the holes and the total number will be calculated after 30 or 60 s depending on the task. Individuals will be given 30 seconds for right hand, left hand and double hand evaluation, while the individual will be given 60 seconds for the evaluation test performed by stacking them one on top of the other with the coordinated movement of both hands, which is called combined movement.
Gross motor skills | 8 weeks
  Box and Block Test:
  The materials required for the test consist of a stopwatch, a wooden box with a centre compartment and 150 wooden cubes. The total duration of the test is 2-5 minutes. Participants will be asked to pass the cubes one by one from one compartment to the other compartment within 60 seconds and the number of cubes will be noted. This test will be applied separately for both extremities.
Gait characteristics | 8 weeks
  10 Metre Walk Test: The 10 Metre Walk Test will be used to determine walking speed. Within the scope of the test, an area of 10 metres will be determined and the time taken to walk this distance will be recorded. A mobile application (OneStep) will be used to record walking speed. The individuals will be asked to walk a distance of 10 metres by placing the phone in the right pocket of their trousers. Time to perform the test, number of steps, step duration, step length, cadence and walking speed values will be recorded.
Dual task performance/Walking | 8 weeks
  10 Metre Walk-Verbal Fluency Test (10MW-VFT): The phone will be placed in the right pocket of the individuals' trousers and they will be asked to say words starting with the letter "A" aloud while walking a distance of 10 metres. The number of steps, step duration, step length, cadence, walking speed, time to perform the test, and the number of correct and incorrectly spoken words will be recorded.
  10 Metre Walk-Serial Subtraction Test: The phone will be placed in the right pocket of the individuals' trousers and while walking a distance of 10 metres, they will be asked to count backwards by subtracting 3 from a randomly selected number between 200-300. The walking characteristics and words will be recorded same as 10MW-VFT.
Dual task performance/Sitting | 8 weeks
  Purdue Pegboard-Verbal Fluency: While performing the Purdue Pegboard test, the patient will be asked to count words starting with the letter 'S' within 30 seconds. The test will be conducted separately for the right and left hand. At the end of the test, the correct answer and the number of sticks will be recorded.
  Purdue Pegboard-Serial Subtraction Test: During the Purdue Pegboard test, individuals will be asked to count backwards by 3 from a number between 300-400 within 30 seconds. The test will be performed separately for the right and left hand. At the end of the test, the correct answer and the number of sticks will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Fatma Bilgin, MSc PT, Principal Investigator — Eastern Mediterranean University; Gözde İyigün, PhD, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Eyalet/Yerleşke, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided